CLINICAL TRIAL: NCT02731417
Title: Acupuncture Treatment for Post-partum Urinary Retention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, wamir, Prof., Rambam Health Care Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0590-15
Record Dates: First submitted 2016-03-06; First posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Urinary retention-group 1 (Experimental): For women with post partum urinary retention designated for experimental treatment.
  Interventions: Other: acupuncture
- Urinary retention-group 2 (Active Comparator): For women with post partum urinary retention designated for current departmental protocol treatment.
  Interventions: Device: Foley catheter

INTERVENTIONS:
Other: acupuncture — Acupuncture for women with post partum urinary retention
  Arms: Urinary retention-group 1
Device: Foley catheter — Foley catheter insertion for women with post partum urinary retention.
  Arms: Urinary retention-group 2

SUMMARY:
There are no set national guidelines for the management of postpartum bladder. There is little evidence on the management of postpartum urinary retention and many hospitals have implemented their own postpartum bladder care protocols.

Acupuncture has been implemented as an alternative course of treatment for urinary retention with reports of spontaneous restoring of micturition in all of the patients. The investigators aimed at examining if acupuncture is a useful tool to treat postpartum urinary retention.

DETAILED DESCRIPTION:
Urinary retention is a common and frustrating complication in women during the immediate postpartum period. Physiologic changes in the bladder that occur during pregnancy predispose patients to develop symptomatic retention of urine during the first hours to days after delivery.

Postpartum urinary retention has a reported incidence ranging from 1.7 to 17.9 percent. Up to 5% of these women may have significant and longer lasting dysfunction, which if not recognised in the early peripartum period, may lead to bladder distension and overflow incontinence with significant long-term bladder dysfunction. Factors associated with postpartum urinary retention include: (1)Nulliparous women. (2) Prolonged labour, especially a prolonged second stage. (3)Assisted/instrumental delivery. (4)Perineal injury. (5)Caesarean section. (6)Regional analgesia.

Treatment begins with supportive measures to enhance the likelihood of micturition, such as ambulation, privacy, and a warm bath. If these measures are not successful, catheterization is usually performed.

There are no set national guidelines for the management of postpartum bladder care as yet. There is little evidence on the management of postpartum urinary retention and many hospitals have implemented their own postpartum bladder care protocols.

Acupuncture has been implemented as an alternative course of treatment for urinary retention in several chinese medical centers over the years with reports of spontaneous restoring of micturition in all of the patients.

A prospective study including all patients with postpartum urinary retention meeting the study criteria will be recruited. All patients will be required to give their informed consent. All patients will undergo a pre-treatment and post-treatment ultrasound recording the residual urine volume.

After the pre-treatment ultrasound acupuncture will be performed according to the following: 1) The points Sanyinjiao (SP 6) and Zusanli (ST 36) on the right side will be punctured 1/5-2 cm deep and moderate stimulation will be applied. 2) The needles will be retained for 30 minutes after achieving Qi and will be manipulated once every 3-5 minutes. After 30 minutes of acupuncture treatment, the patient will have an opportunity to void. If the patient is successful in voiding a post-treatment ultrasound recording the residual urine volume will be performed. If the post-void residual (PVR) urine volume is less than 100 ml acupuncture treatment will be considered a success. If the patient is not successful at voiding during the hour after acupuncture treatment, a post-treatment ultrasound recording the residual urine volume will be performed. If the post-void residual (PVR) urine volume is greater than 100 ml, acupuncture treatment will be considered a failure and the patient will be catheterized.

ELIGIBILITY:
Inclusion Criteria:

* Patients with postpartum urinary retention with either difficulty having voluntary micturition or a post-void residual (PVR) urine volume greater than 100 ml. confirmed by ultrasonography.

Exclusion Criteria:

* Patients with dermatitis over the acupuncture points,
* active urinary tract infection, prior use of anti-cholinergic drugs, cholinergic drugs, and alpha blockers.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
urine residual volume following acupuncture | one hour following acupuncture
  If micturition is achieved within one hour of acupuncture - residual urine volume in bladder is measured by ultrasound (ml).

IPD SHARING:
Plan to Share IPD: Undecided